CLINICAL TRIAL: NCT05118243
Title: Innovative Tools to Produce Legume-based Foods for Increased Consumer Acceptance
Acronym: LeguComf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anne-Maria Pajari, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LeguComf-HY
Record Dates: First submitted 2021-10-08; First posted 2021-11-11 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-masked - neither the researchers or the participants know which cracker they are eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control cracker (Active Comparator): All participants eat control crackers, which contain high amounts of GOS (approx. 5g GOS/daily portion of crackers)
  Interventions: Other: Control cracker
- Enzyme-treated cracker (Active Comparator): All participants eat enzyme-treated crackers, which contain minimal amounts of GOS (less than 1g GOS/daily portion of crackers)
  Interventions: Other: Enzyme-treated cracker

INTERVENTIONS:
Other: Control cracker — The gut symptoms caused by control crackers are studied in IBS persons
  Arms: Control cracker
Other: Enzyme-treated cracker — The gut symptoms caused by enzyme-treated crackers are studied in IBS persons
  Arms: Enzyme-treated cracker

SUMMARY:
The aim of this study is to investigate the effects of enzymatic treatment to reduce GOS (galactooligosaccharides) in legume-based crackers in IBS (irritable bowel syndrome) persons. The crackers are pea-based: the control crackers contain high amounts of GOS, while the enzymatically treated crackers contain a minimal amount of GOS. The participants will eat each type of cracker for three days (daily dose of 12 crackers) and report their gut symptoms (e.g. flatulence, stomach pain, bloating) by using a mobile app. There is a washout period of four days between the different crackers. In addition, the participants will keep food records on the cracker eating days as well as collect five fecal samples during the study. The participants will also report their physical activity and the number of defecations on each day. The study is carried out in a double-blinded crossover setting.

DETAILED DESCRIPTION:
A human intervention study with volunteers suffering from either irritable bowel syndrome (IBS) or functional bloating (FB) will be carried out to investigate the effects of enzymatic treatment of pea-based product on gastrointestinal symptoms and gut microbiota composition as well as hydrogen production due to carbohydrate fermentation. Enzyme-treated product will be compared to a control product.

The aim of the study is to investigate, whether enzyme-treated cracker, compared to a control product, will reduce gastrointestinaI symptoms, or have an impact on fecal microbiome or carbohydrate fermentation measured by breath hydrogen concentration. The effects of eating enzyme-treated crackers on food intake, exercise and stool frequency will also be investigated.

The study is carried out in a randomized, double-blinded, placebo-controlled crossover design. The study includes two 1-week treatment periods with 1-week run-in period before the intervention. Participants (N=35 at the maximum) are adult males and females who meet Rome IV criteria for IBS or FB.

Exclusion criteria will be as follows:

* coeliac disease
* inflammatory bowel disease
* pregnancy or breastfeeding
* antibiotics within the last 3 months
* colonoscopy and preparations for it within 4 weeks

During both treatment weeks each participant will receive three-day portion of either α-galactosidase-treated or control pea-based crackers. The participants will be advised to avoid foods that trigger their gastrointestinaI symptoms and otherwise follow their habitual diets for the whole 3-week study period. They will be asked to report severity of nine gastrointestinaI symptoms, keep food record, collect fecal samples, measure breath hydrogen and report their physical activity as well as stool frequency.

The participants will report their gastrointestinal symptoms throughout the study weeks (twice a day on cracker eating days, once on washout days). Physical activity and stool frequency will also be reported daily. Fecal samples will be collected during the run-in period (at baseline) and on third and seventh day of each treatment week. Breath hydrogen will be measured on second day of both treatment weeks. Nutrient intake and food consumption will be analyzed from 3-day food records during the run-in week and each treatment week (total 9 days). Nutrient intake will be calculated using a new Finnish 'Aromi Diet' software.

ELIGIBILITY:
Inclusion Criteria:

* IBS (Rome IV criteria) or functional bloating
* over 18 years old

Exclusion Criteria:

* IBD (inflammatory bowel disease)
* coeliac disease
* pregnancy or breastfeeding
* antibiotics within the last 3 months
* colonoscopy and preparations for it within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The intensity of stomach pain measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced stomach pain on a scale of zero (no pain at all) to 100 (very intense pain) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of stomach cramps measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced stomach cramps on a scale of zero (no cramps at all) to 100 (very intense cramps) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of bloating measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced bloating on a scale of zero (no bloating) to 100 (very bloated) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of flatulence measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced flatulence on a scale of zero (no flatulence at all) to 100 (very intense flatulence) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of stomach noise measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced stomach noise on a scale of zero (no noise at all) to 100 (very loud noise) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of nausea measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced nausea on a scale of zero (no nausea at all) to 100 (very intense nausea) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of heartburn measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of experienced heartburn on a scale of zero (no heartburn at all) to 100 (very intense heartburn) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of an unpleasant feeling in the upper abdomen or the feeling of feeling full fast related to eating measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of an unpleasant feeling in the upper abdomen or the feeling of feeling full fast related to eating on a scale of zero (no no described unpleasant feeling at all) to 100 (very intense unpleasant feeling) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The intensity of a sudden need to defecate measured by a visual analogue scale | 2 weeks
  Study participants report the intensity of a sudden need to defecate on a scale of zero (no need to defecate at all) to 100 (very intense need to defecate) using a mobile application. The data will be summarized in Excel form and the differences between the treatments will be analyzed statistically.
The composition of gut microbiota analyzed from fecal samples using 16S rRNA amplicon sequencing | 2 weeks
  The composition of gut microbiota is analyzed from fecal samples using 16S rRNA amplicon sequencing and qPCR (quantitative polymerase chain reaction). The differences between the treatments will be analyzed statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maria Pajari, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared